CLINICAL TRIAL: NCT06025149
Title: Open, Prospective, Multicenter Study of the Safety and Efficacy of "UniLine" Epoxy-treated Prosthesis Made From Xenopericardium in the Treatment of Isolated Aortic and Mitral Valve Diseases
Brief Title: The Study on the Use of "UniLine" Bioprosthesis in the Treatment of Isolated Aortic and Mitral Valve Diseases
Acronym: Uniline
Status: Recruiting | Type: Observational
Sponsor: Closed Joint-Stock Company NeoCor (Other)
Collaborators: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other); CT Medical Limited Liability Company (Unknown)
Responsible Party: Sponsor
Other Study IDs: UniLine
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Aortic Valve Disease; Mitral Valve Disease
Keywords: UniLine biological prosthesis; Acquired valve disease; Acquired aortic valve disease; Acquired mitral valve disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this open, prospective, multicenter study is analyze long-term outcomes of aortic/mitral valve replacement using the "UniLine" bioprosthesis in patients with acquired aortic or mitral valve diseases.

Main research objectives:

To analyze long-term (up to 12 years) outcome of aortic or mitral valve replacement using the "UniLine" bioprosthesis.

To study the hemodynamic characteristics of normally functioning "UniLine " prostheses in the mitral or aortic valve position based on the transthoracic echocardiography data.

To assess the number, type, time frames of dysfunctions of UniLine bioprostheses and the results of their treatment.

To analyze the frequency of major serious adverse events associated with the "UniLine" bioprosthesis or procedure.

DETAILED DESCRIPTION:
Acquired heart diseases (AHDs) remain one of the most frequent causes of cardiac mortality and disability. In Russia, this kind of disease accounts for 7 to 25 % of all cardiovascular diseases, and is third most common cause of heart failure.

Heart valve replacement using a prosthetic heart valve remains the main and most effective method of treatment of AHDs. In Russia, AHDs are treated in more than 40 subjects by specialists from 92 medical institutions. Valve replacements, being high-tech methods of treatment, most effectively prolong the life of patients. Timely correction of AHD allows 75-95 % of patients to return to a normal lifestyle.

The aim of this study is to evaluate the safety and effectiveness of the "UniLine" epoxy-treated bioprosthesis in the treatment of isolated mitral or aortic heart valve diseases.

The expected clinical benefit involves the treatment of valvular disease with restoration of intracardiac hemodynamics during implantation of the "UniLine " bioprosthetic valve, followed by remodeling of the heart chambers, which should lead to an improvement in heart function and quality of life of the patient.

The expected risks are associated with taking anticoagulant therapy during the first three months after implantation, or as a result of prolonged anticoagulant therapy, in the presence of concomitant rhythm disturbances, and consist in the possibility of hemorrhagic or thromboembolic complications.

ELIGIBILITY:
Inclusion Criteria:

1. Provided informed consent to participate in the study.
2. Must be aged 18 years and older.
3. Patients with isolated acquired mitral or aortic valve disease.
4. No prior heart valve replacement, current replacement must be planned (not conducted in an urgent/ emergency manner), using the "UniLine" biological prosthesis made from xenopericardium.
5. Patient must be able to visit the Research Center.

Exclusion Criteria:

1. Mechanical or biological prosthesis in another position. Patients with tricuspid valve repair may be included in the study.
2. Prior heart valve replacement.
3. Concomitant interventions on the heart (coronary artery bypass grafting, coronary heart disease treatment, surgical reconstruction of a left ventricular aneurysm) and thoracic aorta.
4. Patients with cancer in history.
5. Patients with musculoskeletal conditions with severe movement disorders and diseases of the central nervous system, accompanied by cognitive disorders (disorientation, inability to independently reach the destination).
6. Acute or subacute stages of infective endocarditis.
7. Class IV heart failure according to the New York Heart Association Functional Classification with ongoing therapy, left ventricular ejection fraction less than 40%, myocardial infarction less than 90 days old, angina pectoris grade 4.
8. The presence of severe somatic, neurological, mental and infectious diseases that worsen the prognosis of long-term survival: tuberculosis, human immunodeficiency virus, Alzheimer's disease, epilepsy, chronic kidney disease stage 3b (Glomerular Filtration Rate less than 30 mL/ min / 1.73 m²), chronic lung diseases requiring constant intake of corticosteroids and bronchodilators, multifocal atherosclerosis (grade 3 chronic lower limb ischemia, stenosis of the carotid arteries more than 50%, prior and planned interventions on the abdominal aorta, carotid arteries or arteries of the lower extremities).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As part of these clinical trials (studies), the use of comparison groups is not planned.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-09-09 (Estimated); Study Completion 2035-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the Bioprosthetic Valve | 12 years since the replacement surgery
  Safety of using the bioprosthesis is defined as the absence of major adverse events related to the device or procedure, assessed using the following clinical phenomena:
  1. Fatal outcome: a) all-cause death; b) related to cardiovascular diseases; c) related to the dysfunction of the prosthesis.
  2. Life-threatening bleeding.
  3. Any dysfunction associated with the bioprosthesis (stenosis, regurgitation), migration of the device, thrombosis or other complication requiring surgical intervention.
  4. Any dysfunction associated with the bioprosthesis that does not require surgical intervention.
  5. Myocardial infarction (or stroke) or progression of a chronic form of ischemia requiring percutaneous coronary intervention or coronary artery bypass graft surgery
  6. Stroke
Long-Term Durability of the Bioprosthetic Valve | 12 years since the replacement surgery
  It will be evaluated by measuring the hemodynamic characteristics of the prosthetic valve, assessed by echocardiography: maximum, average gradients and effective orifice area (absolute and indexed values).

SECONDARY OUTCOMES:
Hemodynamic characteristics of the Bioprosthetic Valve | 12 years since the replacement surgery
  They will be assessed by using echocardiography: maximum, average gradients and effective orifice area (absolute and indexed values).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bogachev-Prokofiev, MD, PhD, Principal Investigator — National Medical Research Center named after Academician E.N. Meshalkin; Alexey Evtushenko, MD, PhD, Principal Investigator — Research Institute for Complex Issues of Cardiovascular Diseases
Locations (1):
- Research Institute for Complex Problems of Cardiovascular Diseases, Russia, Kemerovo, Kemerovo Oblast, Russia